CLINICAL TRIAL: NCT01511406
Title: Does Cognitive Behavioral Therapy Improve Depressive Symptoms and Self-Esteem in Patients With a First Episode Psychosis? A Randomized Controlled Study
Brief Title: Cognitive Behavioral Therapy for Patients With an Early Psychosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Stiftelsen Helse og Rehabilitering (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CBT2011
Record Dates: First submitted 2011-12-27; First posted 2012-01-18 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Psychosis; Schizophrenia; Depressive Symptoms; Self-esteem
Keywords: Psychosis; Schizophrenia; Cognitive behavioral therapy; Self esteem; Depression
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- cognitive behavioral therapy (Experimental): Cognitive behavioral therapy up to 26 sessions
  Interventions: Behavioral: cognitive behavioral therapy

INTERVENTIONS:
Behavioral: cognitive behavioral therapy — Patients allocated to the treatment arm will receive up to 26 sessions of cognitive behavioral therapy
  Other Names: CBT

SUMMARY:
The purpose of the present study is to examine whether cognitive behavior therapy will reduce depressive symptoms and increase self-esteem for patients with a first episode psychosis.

DETAILED DESCRIPTION:
A growing body of evidence supports the use of Cognitive Behavioural Therapy (CBT) for the treatment of schizophrenia. The strength of evidence is especially strong for patients with persistent hallucinations and delusions. As it comes to the effect of CBT for patients with a first episode psychosis the picture is more unclear. The main reason is probably that the CBT interventions to a less extent have been adjusted to fit first episode psychosis patients. The main problems for patients with a first episode psychosis (FEP) is rarely persistent hallucinations and delusions but they struggle with social anxiety, depression, alcohol and drug abuse and low self esteem. Forthcoming studies examining the effect of CBT for patients with a first episode psychosis should aim to have a focus on these symptoms.

The main aim of the present study is to examine whether CBT has any effect on depressive symptoms and self-esteem in patients with a FEP.

The study will include patients with a first episode psychosis with Axis-I DSM IV diagnosis of schizophrenia, schizoaffective disorder, delusional disorder, and psychosis not otherwise specified. To be included in the study the patients should meet the criteria of an affective episode the last year or have a score on Calgary Depression of Schizophrenia Scale above four. Patients are randomly selected to either a treatment group or a control (placebo) group. The aim is to include 30 patients in each group. Patients in the treatment group will receive a manual-based CBT intervention comprising up to 26 sessions during a six months period. The control group will receive treatment as usual (TAU).

The patients are assessed before the entry of the study and after 6 months (end of treatment). Moreover they will be assessed after 9 months of ending therapy.

Hypothesis:

In this study we hypothesize that

* patients receiving CBT will have less depressive symptoms than TAU-patients at the and of treatment and at six months follow up
* CBT-patients will demonstrate a better improvement in their self-esteem than TAU-patients at the end of treatment and at six months follow up.

To our knowledge, no previous studies have examined outcome after CBT treatment with regards to depressive symptoms and self-esteem. Furthermore, this is the first randomized controlled study in Norway of CBT among patients with a FEP.

ELIGIBILITY:
Inclusion Criteria:

* Participants are eligible for the study if they are diagnosed with a psychotic disorder or bipolar disorder with psychosis according to DSM-IV (i.e. schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder or psychosis NOS
* Aged between 18-65 years
* Are capable of giving a written consent to participate in the study.

Exclusion Criteria:

* A history of head injury, neurological disorders, developmental disorders, and all episodes of psychosis being judged as substance-induced rather than a primary episode of a psychotic disorder.
* Being in treatment for more than five years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Calgary Depression rating Scale for Schizophrenia (CDSS) | up to nine months after end of intervention
  Measure depressive symptoms for patients with a psychosis

SECONDARY OUTCOMES:
Rosenberg Self Esteem Scale | up to nine months after end of intervention
  Measure the level of self esteem among patients with a psychosis

CONTACTS AND LOCATIONS:
Overall Officials: Jan I Røssberg, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Sonmez N, Romm KL, Ostefjells T, Grande M, Jensen LH, Hummelen B, Tesli M, Melle I, Rossberg JI. Cognitive behavior therapy in early psychosis with a focus on depression and low self-esteem: A randomized controlled trial. Compr Psychiatry. 2020 Feb;97:152157. doi: 10.1016/j.comppsych.2019.152157. Epub 2019 Dec 26. PMID 31935529